CLINICAL TRIAL: NCT04486937
Title: Sc10914 Monotherapy for Metastatic Castration Resistant Prostate Cancer Patients With Germ and / or Somatic BRCA Mutation: a Single Arm, Multicenter Clinical Tria
Brief Title: SC10914 Monotherapy for the mCRPC With g/s BRCA Mutation
Acronym: mCRPC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QF-SC10914-202
Record Dates: First submitted 2020-07-20; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SC10914 (Experimental): 400mg TID，oral admination on an fasting state
  Interventions: Drug: S410914 tablet

INTERVENTIONS:
Drug: S410914 tablet — S410914 tablet

SUMMARY:
This study is a multicenter, single arm phase I / II clinical study in mCRPC subjects who failed to receive docetaxel chemotherapy, abitolone acetate and / or enzalutamide (including its analogues) for the treatment of BRCA mutations in germ cells and / or somatic cells.

DETAILED DESCRIPTION:
The subjects oral administration sc10914 tablets 400mg on an empty stomach, three times a day, for 28 consecutive days as a treatment cycle, until disease progression (PD) (according to Recist1.1 and the adjusted PCWG3 standard, the subjects met the imaging [CT / MRI / bone scan] PD standard) or the toxicity was intolerable.

The study is divided into two stages: in the first stage,enrolled 36 patients whose response can be evaluated, if there are at least 7 cases of objective remission (CR or PR), the second stage is allowed, otherwise the study will be stopped; in the second stage, the number of subjects whose response can be evaluated is planned to continue to be enrolled to 70 cases（stage 1 and stage 2）.

ELIGIBILITY:
Inclusion Criteria:

1. Signing informed consent voluntarily;
2. Prostate cancer confirmed by histology or cytology;
3. Metastatic lesions proved by imaging (CT / MRI / bone scan);
4. At least one measurable lesion in accordance with recist1.1;
5. deleterious or suspected deleterious germline and/or somatic BRCA-mutated (g/sBRCAm)
6. ECOG≤2；
7. The expected survival time was more than 3 months;
8. Serum testosterone levels ≤ 50 ng/dL (≤ 1.75 nmol/L) at screening.
9. Subjects without prior surgical castration must be currently taking and willing to continue luteinizing hormone-releasing hormone (LHRH) analog (agonist or antagonist) therapy throughout the duration of study treatment.

9.Subjects must have progressed on prior NHA (e.g. abiraterone acetate and/or enzalutamide) for the treatment of mCRPC. 10.Subjects must have progressed on prior chemotherapy with docetaxel for the treatment of mCRPC.

Exclusion Criteria:

1. Any previous treatment with PARP inhibitor
2. Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors. The required washout period prior to starting olaparib is 2 weeks or 5 half-life.
3. Subjects with known brain metastases.
4. Major surgery within 2 weeks of starting study treatment and subjects must have recovered from any effects of any major surgery
5. Subjects unable to swallow orally administered medication and subjects with gastrointestinal disorders likely to interfere with Absorption, distribution, metabolism and excretion of the study
6. Immunocompromised subjects, e.g., subjects who are known to be serologically positive for human immunodeficiency virus (HIV)
7. Subjects with a known hypersensitivity to SC10914 or any of the excipients of the product
8. Subjects with known active hepatitis (i.e. Hepatitis B or C)
9. Subjects with not enough organ functional reserve at baseline, which met at least one of the following criteria：

   1. ANC<1.5×109/L；
   2. PLT<100×109/L；
   3. Hb<100g/L；
   4. TBIL>1.5×ULN；
   5. ALT、AST>2.5×ULN unless liver metastases are present in which case they must be > 5×ULN；
   6. Cr >1.5×ULN。
10. Subjects who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

    1. Baseline QT interval corrected for heart rate (HR) using Fridericia's formula >500 msec or congenital long QT syndrome;
    2. Left ventricular ejection fraction (LVEF) <50% assessed by echocardiogram;
    3. Other clinically significant heart disease such as congestive heart failure NYHA Class IV and requiring heart transplant
11. Severe bone injury caused by tumor bone metastases as judged by the researchers, including severe bone pain due to poor control, pathological fracture of important parts or spinal cord compression occurred or expected to occur in the near future in the last 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | up to 100 weeks (estimated)
  assessed by the independent imaging assessment committee (recist1.1)

SECONDARY OUTCOMES:
PFS | up to 100 weeks (estimated)
Disease control rate (DCR), duration of response (DOR), time to tumor progression (TTP) | up to 100 weeks (estimated)
  evaluated according to recist1.1 and adjusted pcwg3 criteria
overall survival (OS) | up to 100 weeks (estimated)
  evaluated according to recist1.1 and adjusted pcwg3 criteria

IPD SHARING:
Plan to Share IPD: No